CLINICAL TRIAL: NCT04858243
Title: Engaging Men Through HIV Self-Testing With Differentiated Care to Improve ART Initiation and Viral Suppression Among Men in Malawi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: Partners in Hope, Inc. (Industry); Medical University of South Carolina (Other); Charles University, Czech Republic (Other); University of Cape Town (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Thomas J. Coates, Director of University of California Global Health Institute, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH122308 (NIH); R01MH122308-01A1 (NIH)
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Hiv
Keywords: HIV; Men; HIV Self-Testing; ART Initiation; ART Retention; Home-Based care; Antiretroviral Therapy; Viral Suppression; Sub-Saharan Africa; Malawi
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facility-Based ART (Active Comparator): Men escorted to nearest health facility for ART initiation and continuation.
  Interventions: Other: Facility-Based ART
- Home-Based ART (Experimental): Home-based ART initiation and continuation provided for 3-months.
  Interventions: Other: Home-Based ART

INTERVENTIONS:
Other: Home-Based ART — Community-based male-specific counseling followed by home-based ART initiation (or at any location that is convenient for participants) and home-based ART continuation for a 3-month period, followed by linkage to a local health facility for further ART continuation.
  Arms: Home-Based ART
Other: Facility-Based ART — Community-based male-specific counseling followed by linkage to a local health facility for ART initiation and continuation.
  Arms: Facility-Based ART

SUMMARY:
Men in sub-Saharan Africa who test HIV-positive continue to have poor ART initiation and retention outcomes. The proposed project will test a home-based ART intervention for men who are living with HIV compared to facility-based ART. Findings will provide essential information on how to best reach men across the testing and treatment continuum, a critical step to curbing the HIV epidemic.

DETAILED DESCRIPTION:
Background: Men in sub-Saharan Africa are less likely than women to use HIV services. HIV testing strategies have dramatically improved for men through HIV self-testing (HIVST) and other male-focused strategies, but men who are identified as living with HIV are still less likely than women to initiate ART or remain in care, particularly within the first several months after initiation. In Malawi, men represent only 31% of new ART initiates2 - and men on ART are more likely than women to be lost to follow up (LTFU) at all time intervals of care than women. Men's absence from care is concerning not only for their own health, but also for the health of girls and young women who continue to be infected at unacceptably high rates. Offering ART at home or other locations convenient for men (i.e., home-based ART) for a brief period of time may help men overcome barriers related to facility-based treatment, develop coping strategies for ART engagement, and better engage in facility-based services over the long-term. In this study we will assess the impact of hbART by comparing two arms:

Facility-Based ART (fbART arm): community-based male-specific counseling followed by linkage to a local health facility for ART initiation and continuation.

Home-Based ART (hbART arm): community-based male-specific counseling followed by home-based ART initiation (or at any location that is convenient for participants) and home-based ART continuation for a 3-month period, followed by linkage to a local health facility for further ART continuation.

Objective: Our primary objective is to compare the impact of home-based ART against standard of care for ART initiation and retention among men identified as HIV-positive through HIVST in Malawi. Our specific Aims are:

Aim 1. Test the effectiveness of hbART versus fbART on ART initiation and 6-month viral suppression among men living with HIV.

Aim 2. Identify predictors of ART initiation and 6-month viral suppression in the hbART arm

Aim 3. Determine the cost-effectiveness and scalability of hbART at a national level.

Methods: We will perform an individually randomized control trial with 820 HIV-positive men who have not yet initiated ART and a subset of 110 of their female partners. Men will be individually randomized 1:1 to one of the two intervention arms described above and will be enrolled in the study for 18-months or until 12-month retention (secondary outcome) can be measured, whichever comes first. The study will be performed at 10 health facilities supported by Partners in Hope (PIH). Data collection will include baseline and follow-up surveys at 2-, 4-, and 7-months, as well as medical charter reviews for men at 2-, 4-, 7-, and 13-months after study enrollment. Qualitative interviews will be conducted with a subset of men and women to understand perceptions of the intervention and experiences with ART engagement, and cost data from a provider perspective will be collected for a cost analysis of each arm.

Anticipated results: Findings will establish the effectiveness of home-based ART among men living with HIV who have not yet engaged in treatment, and can directly inform HIV programs throughout the region. Findings will also help us assess if short-term home-based ART is sufficient to engage men in long-term facility-based care, or if additional, more resource-intensive services are needed, such as major changes to the structure of facility-based ART.

ELIGIBILITY:
Female Partner Inclusion Criteria:

* Male partner ≥15 years of age
* No reported interpersonal violence (IPV) as defined by World Health Organization (WHO) with the above male partner in the past 12-months
* Male partner ever tested HIV-positive
* Male partner not currently engaged in ART services, defined as:

  * Tested HIV-positive ≥14 days and not on ART ≥14 days after testing HIV- positive;
  * ≥14 days late for the first four-week follow up appointment; or
  * Initiated ART but ≥60 days late for last ART appointment;
  * Male partner living inside the facility catchment area (defined as any area that Healthcare Workers (HCWs) from the study facility routinely visit for tracing purposes)

Female Partner Exclusion Criteria:

* Male partner <15 years of age
* Reported interpersonal violence (IPV) as defined by WHO with the above male partner in the past 12-months
* Male partner never tested HIV positive
* Male partner tested HIV-positive <14 days ago
* Male partner currently engaged in ART services, defined as:

  * Initiated ART <14 days late for the first four-week follow up appointment
  * Initiated ART and <60 days late for last ART appointment
  * Male partner living outside the facility catchment area (defined as any area that HCWs from the study facility routinely visit for tracing purposes)

Men Living with HIV Inclusion Criteria:

* ≥15 years of age
* Tested HIV positive using Ministry of Health standard algorithm (Determine + Unigold)
* Not currently engaged in ART services, defined as:

  * Tested HIV-positive ≥14 days and not on ART ≥14 days after testing HIV-positive;
  * ≥14 days late for the first four-week follow up appointment; or
  * Initiated ART but ≥60 days late for last ART appointment;
  * Has not taken ART in the past 7-days, as indicated by a point of care (POC) urine assay
  * Living inside the facility catchment area (defined as any area that HCWs from the study facility routinely visit for tracing purposes)

Men Living with HIV Exclusion Criteria:

* <15 years of age
* Never tested HIV positive using Ministry of Health standard algorithm (Determine + Unigold)
* Tested HIV-positive <14 days ago
* Currently engaged in ART services, defined as:

  * Initiated ART
  * <14 days late for the first four-week follow up appointment
  * Initiated ART and <60 days late for last ART appointment
  * Has taken ART in the past 7-days, as indicated by a point of care (POC) urine assay
  * Living outside the facility catchment area (defined as any area that HCWs from the study facility routinely visit for tracing purposes)

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 930 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
6-month viral suppression among men living with HIV | 12 months
  Proportion of HIV-positive men tested HIV-positive who have an undetectable viral load 6-months after initiating ART (a maximum of 12-months after enrolling in the study). Sourced by medical chart reviews.

SECONDARY OUTCOMES:
ART Initiation | 6 months
  Proportion of HIV-positive male partners tested HIV-positive who initiate ART within 6-months of enrolling in the study. Sourced by medical chart reviews.
ART Retention | 18 months
  Proportion of male partners who initiate and have never been >60 days late for ART within the first 12-months after treatment initiation (max 18 months after enrolment). Sourced by medical chart reviews.
Proportion of female clients and men who self-report at least one adverse event | 18 months
  Self-report of adverse events (IPV, unwanted disclosure, end of relationship) from female ART client and men (unwanted disclosure) enrolled in the study. Source is follow-up surveys.

CONTACTS AND LOCATIONS:
Locations (1):
- Partners in Hope, Lilongwe, Malawi

REFERENCES:
- [Derived] Hubbard J, Mphande M, Robson I, Balakasi K, Phiri K, Chikuse E, Thorp M, Phiri S, Choko AT, Cornell M, Coates T, Dovel K. Core components of male-specific person-centred HIV care: a qualitative analysis from client and healthcare worker perspectives in Malawi. BMJ Public Health. 2024 Dec 22;2(2):e001100. doi: 10.1136/bmjph-2024-001100. eCollection 2024 Dec. PMID 40018627
- [Derived] Holland KN, Hubbard J, Mphande M, Robson I, Phiri K, Onoya D, Chikuse E, Dovel K, Choko A. Implementation of Male-Specific Motivational Interviewing in Malawi: An Assessment of Intervention Fidelity and Barriers to Scale-Up. medRxiv [Preprint]. 2024 Sep 26:2024.09.24.24314326. doi: 10.1101/2024.09.24.24314326. PMID 39399024
- [Derived] Choko AT, Coates TJ, Mphande M, Balakasi K, Robson I, Phiri K, Phiri S, Kulich M, Sweat M, Cornell M, Hoffman RM, Dovel K. Engaging men through HIV self-testing with differentiated care to improve ART initiation and viral suppression among men in Malawi (ENGAGE): A study protocol for a randomized control trial. PLoS One. 2023 Feb 24;18(2):e0281472. doi: 10.1371/journal.pone.0281472. eCollection 2023. PMID 36827327